CLINICAL TRIAL: NCT06781606
Title: Pilot Study of PEnile TRAnsplantation - Vascularized Composite Allografts
Acronym: PETRA-VCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: French Association of Urology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL22_0906; 2024-A02180-47 (Other: ID-RCB)
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Adults with Traumatic Penile Severe Defects; Congenital Penile Defects; Micropenis
Keywords: Penile transplatation; Vascularized Composite Allografts; Allotransplantation; En bloc harvesting; urinary function; sexual function; self-image
MeSH Terms: conditions — Penis agenesis | interventions — Penile Transplantation

STUDY DESIGN:
Intervention Model Description: Prospective, multicentric, non-randomized, pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Penile transplantation (Experimental)
  Interventions: Procedure: Penile transplantation

INTERVENTIONS:
Procedure: Penile transplantation — The penile transplantation will take place at the Edouard Herriot hospital, part of the Hospices Civils de Lyon. It will be carried out on the same day or the day after the harvesting depending on the timing of the harvesting.

SUMMARY:
Penile transplantation (PT) has recently emerged as an option for penile reconstruction and has shown encouraging outcomes at the international level with two ongoing PT program (US, South Africa). Emergence of such option has been possible thanks to the development of vascularized composite allotransplantation and because of the important limitations of autologous reconstruction (phalloplasty). Feasibility has already been proven, but the surgical management remains in its infancy and has never been tested at a European level. Furthermore, the balance between functional improvement and immunosuppressive risk still needs to be enlightened.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years and ≤ 60 years
* Patient with traumatic penile severe defects (amputation), or congenital penile defects (micropenis)
* ASA ≤ 2
* NYHA ≤ 1
* Creatinine clearance > 60 mL/min (CKD-EPI)
* Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Informed consent signed to participate to the study

Exclusion Criteria:

* Gender incongruence
* Congenital penile defects resulting from exstrophy/epispadias
* Penile malformation due to selh-half/self-amputation
* Amputation for penile cancer
* Other types of malignancy in remission for less than 5 years
* Progressive malignant tumor
* Presenting hepatitis B, hepatitis C, or HIV infection not controlled by appropriate anti-viral therapy
* Uncontrolled arterial hypertension
* Moderate renal failure : glomerular filtration rate of less than 60 mL/min per 1.73 m2
* EBV sero-negative recipient with EBV sero-positive graft, due to the risk of lymphoma
* Non controlled chronic infection
* Malignancy, Connective tissue disease
* Amyloidosis
* Unbalanced diabetes
* Patient with a contraindication to performing an MRI examination
* Contra-indication of Thymoglobuline: Hypersensitivity to rabbit proteins or to any of the excipients of Thymoglobuline, acute or chronic infections that contraindicate any additional immunosuppression,
* Contra-inducation of tacrolimus: Hypersensitivity to tacrolimus or others macrolides, or any of the excipients of PROGRAF,
* Contra-indication of Mycophenolate mofetil: in patients with hypersensitivity to mycophenolate mofetil, mycophenolic acid or any of the excipients, Hypersensitivity reactions to mycophenolate mofetil;
* History of major psychiatric disorders < 3 years (psychotic disorders, severe substance abuse, severe personality disorders) or persons under psychiatric care ;
* Person deprived of their liberty by a judicial or administrative decision ;
* Person admitted to a health or social institution for purposes other than research
* Adult subjects to a legal protection measure (guardianship, curatorship)
* Person not affiliated to a social security scheme of beneficiaries of a similar scheme

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete functional evaluation | 24 months
  Complete functional evaluation after penile transplantation, including the different function of the phallus : Urinary function (uroflowmetry, post-voiding residual voluma and Urinary Symptom Profile (USP®) );
Complete functional evaluation | 24 months
  Complete functional evaluation after penile transplantation, including the different function of the phallus : sexual function (penile doppler ultrasonography, nocturnal penile tumescence, Erection Hardness Score (EHS) and the International Index of Erectile Function (IIEF)).
Complete functional evaluation | 24 months
  Complete functional evaluation after penile transplantation, including the different function of the phallus : aesthetics and self-image (Rosenberg scale, Male Genital Self-image Scale (MGSIS), Self Esteem and Relationship questionnaire (SEAR))

SECONDARY OUTCOMES:
Complete functional evaluation | Preoperatively, 6 months and 12 months
  Complete functional evaluation after penile transplantation, including the different function of the phallus : Urinary function (uroflowmetry, post-voiding residual voluma and Urinary Symptom Profile (USP®) );
Complete functional evaluation | Preoperatively, 6 months and 12 months
  Complete functional evaluation after penile transplantation, including the different function of the phallus : sexual function (penile doppler ultrasonography, nocturnal penile tumescence, Erection Hardness Score (EHS) and the International Index of Erectile Function (IIEF))
Complete functional evaluation | Preoperatively, 6 months and 12 months
  Complete functional evaluation after penile transplantation, including the different function of the phallus : aesthetics and self-image (Rosenberg scale, Male Genital Self-Image Scale (MGSIS), Self Esteem and Relationship questionnaire (SEAR))
Postoperative complications | up to 60 months
  Any surgical complications which occur in the first three months post transplantation will be collected , they will be assessed according to their cause and level of severity (Clavien-Dindo Classification). Infectious and metabolic complications, side effects of immunosuppression including renal function, New Onset Diabetes After Transplantation (NODAT), infection, incidence of post-transplant malignancy will be collected throughout the study from blood tests and ECBU. Acute organ rejection evaluation will be evaluated by allograft biopsy (lymphocytic infiltrate, apoptosis, artery endothelialitis)
Qualitive evaluation | Preoperatively, 6 months, 12 months and 24 months
  Semi-structured patient interviews will be performed. The preoperative interview will investigate the functional aspects of urination and sexuality when suffering from penile defect. A specific interest will be given to the expectations of the patient and foreseen benefit of PT. The appropriation and the experience of allotransplantation will be explored along with the different functionnal domains.
Health-economic evaluation | 24 months
  The cost per penile transplantation procedure including transplant preparation will be estimated from the hospital perspective. Moreover the quantity of resources consumed and the total penile transplantation cost per patient including post-transplantation cost follow-up cost will be assessed from the health care system perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Neuville, Doctor, Principal Investigator — Service d'urologie Hôpital Lyon Sud
Locations (9):
- France (9):
  - Service d'urologie, andrologie et transplantation rénale Groupe hospitalier Pellegrin Tripode CHU Bordeaux, Bordeaux
  - Service d'urologie, andrologie et transplantation rénale Hôpital Huriez CHRU Lille, Lille
  - Service d'urologie, chirurgie de la transplantation Hôpital Edouard Herriot Hospices Civils de Lyon, Lyon
  - Service de chirurgie urologique et transplantation rénale AP-HM Hôpital de la Conception, Marseille
  - Service de chirurgie des brûlés, plastique, reconstructrice et esthétique Polyclinique Saint Roch, Montpellier
  - Service néphrologie - soins intensifs - dialyse et transplantation CHU de Montpellier, Montpellier
  - Service d'urologie Hôpital Lyon Sud, Pierre-Bénite
  - Service d'urologie Hôpital Foch, Suresnes
  - Département d'urologie, andrologie et transplantation rénale Hôpital Rangueil CHU de Toulouse, Toulouse